CLINICAL TRIAL: NCT03375541
Title: Benefits of Drug Risk Aversion Calculation to Multiple Sclerosis Drug Choice and Patient Self-efficacy
Brief Title: Drug Risk Aversion Calculator Use to Facilitate MS Patient Self-efficacy
Acronym: DRAC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinical workflow was too high
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00081429
Record Dates: First submitted 2017-12-08; First posted 2017-12-18 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Natural discussion of disease modifier selection conducted without augmentation by risk aversion calculator
- Calculator (Experimental): Natural discussion of disease modifier selection conducted with augmentation by risk aversion calculator
  Interventions: Other: Risk Aversion Calculator

INTERVENTIONS:
Other: Risk Aversion Calculator — The calculator asks the participant to rate their level of aversion to having a set list of potential medication side effects (0 = no concern; 1 = mild concern; 2 = moderate concern; 3 = moderate to severe concern; 4 = severe concern)
  Arms: Calculator

SUMMARY:
The investigators seek to determine if the use of a Side Effect Aversion Calculator helps patients with multiple sclerosis (MS) more comfortably and rapidly identify the disease modifying drug (DMD) that is best suited for the patient.

DETAILED DESCRIPTION:
Settling into the use of a multiple sclerosis disease modifying drug (DMD) can seem like taking an important final examination, consisting of a single multiple choice question with 16 equally appropriate responses, having months or even years to second-guess your choice, and then getting a grade but never being told the correct answer.

Making the choice between these options can be overwhelming, leaving patients feeling both disempowered and depersonalized in the decision-making process.

In order to allow a better, more personalized, decision-making process the investigators introduce a side effect aversion calculator, which takes a patient's individual side effect aversion profile into consideration when discussing the start of a new disease modifier (initial drug, or drug switch). Subjects will be multiple sclerosis patients who have a provider-identified need for DMD initiation or DMD switch and receive their care at Duke. Recruitment goal is 100 subjects. Those randomized to "calculator arms" will be reminded that the purpose of the calculator is to facilitate the DMD choice discussion, NOT make the decision. Subjects asked to rate level of concern over adverse events (AEs) across all DMDs. Calculator multiplies subject response by the prevalence reported within DMD prescribing information. Sum of these weighted scores reveals a DMD's Total Aversion score and medication ranking by patient's specific side effect aversion profile, therefore framing discussion. Enrollment visit concludes with survey designed to collect MS clinical history, MS symptoms, medication history, medication adherence and self-efficacy. This same survey is conducted prior to subsequent three clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Be able to read and speak English
* Be currently treated or starting treatment with an MS disease modifying medication

Exclusion Criteria:

* All of the inclusion criteria must be met. If they cannot be met, then they are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Disease Self-efficacy | Baseline and then at the conclusion of the initial 1 day visit
  Degree of change over time in a person's judgement of how well one can execute courses of action required to manage multiple sclerosis

SECONDARY OUTCOMES:
Time to new medication start | 6 months
  The amount of time (in days) from initial treatment discussion to treatment start
Medication adherence | At enrollment and at each subsequent visit for one year
  The percentage of all prescribed doses of a medication that a patient takes
Change from Baseline Disease Self-efficacy at 6 months | At enrollment and at 6 months post-visit
  Degree of change over time in a person's judgement of how well one can execute courses of action required to manage multiple sclerosis
Change from Baseline Disease Self-efficacy at 12 months | At enrollment and at 12 months post-visit
  Degree of change over time in a person's judgement of how well one can execute courses of action required to manage multiple sclerosis

CONTACTS AND LOCATIONS:
Overall Officials: Fletcher Hartsell, MD MPH, Principal Investigator — Duke University